CLINICAL TRIAL: NCT06082843
Title: Randomised, Double-blind, Placebo-controlled and Parallel Group Trial to Investigate the Effects of One Dose (Up-titration to a Fixed Dose Regimen) of Oral BI 685509 on Portal Hypertension After 8 Weeks Treatment in Patients With Clinically Significant Portal Hypertension (CSPH) in Decompensated Cirrhosis After Their First Decompensation Event, Who Are Stabilized CTP 5-7
Brief Title: A Study to Test Whether Avenciguat Helps People With Liver Cirrhosis and High Blood Pressure in the Portal Vein (Main Vessel Going to the Liver) Who Had Bleeding in the Esophagus or Fluid Accumulation in the Belly
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Company decision
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 1366-0055; 2023-506083-13-00 (Registry Identifier: CTIS)
Record Dates: First submitted 2023-10-09; First posted 2023-10-13 (Actual); Results first posted 2025-06-12 (Actual); Last update posted 2025-06-12 (Actual); Status verified 2025-05

CONDITIONS: Hypertension, Portal; Liver Cirrhosis
MeSH Terms: conditions — Hypertension, Portal; Liver Cirrhosis

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Placebo (Placebo Comparator): Participants with stabilized decompensated cirrhosis due to non-cholestatic liver disease, following their first decompensation event, received 1 milligram (mg), 2 mg, or 3 mg film-coated tablets of placebo-matching avenciguat (BI 685509) orally twice daily (bid). Participants started the treatment with a 1 mg film-coated tablet of placebo-matching avenciguat administered bid. One week later (Visit 3), the dosage was increased to 2 mg film-coated tablets bid, and after another week, participants started on 3 mg film-coated tablet bid (Visit 4), which was maintained for the rest of the treatment.
  Interventions: Drug: Placebo
- Avenciguat (Experimental): Participants with stabilized decompensated cirrhosis due to non-cholestatic liver disease, following their first decompensation event, received 1 milligram (mg), 2 mg, or 3 mg film-coated tablets of avenciguat (BI 685509) orally twice daily (bid), up to a total dose of 6 milligrams (mg). The treatment period began (Visit 2) with a 1 mg film-coated tablet of avenciguat administered bid. If the dose was well-tolerated, it was increased to 2 mg film-coated tablets bid after one week (Visit 3), followed by an increase to the maintenance dose of 3 mg film-coated tablet one week later (Visit 4). If the maintenance dose of avenciguat was not well-tolerated, it was reduced, with the participants remaining on the highest tolerated dose for the rest of the treatment period.
  Interventions: Drug: Avenciguat

INTERVENTIONS:
Drug: Placebo — Placebo-matching Avenciguat
  Arms: Placebo
Drug: Avenciguat — 1 millligram (mg), 2 mg, or 3 mg film-coated tablet
  Other Names: BI 685509
  Arms: Avenciguat

SUMMARY:
This study is open to adults with advanced liver cirrhosis caused by hepatitis B, hepatitis C, alcohol-related liver disease, non-alcoholic steatohepatitis or other causes. People can join the study if they have high blood pressure in the portal vein (main vessel going to the liver) and bleeding in the esophagus or fluid accumulation in the belly. The purpose of this study is to find out whether a medicine called avenciguat helps people with this condition.

Participants are put into 2 groups by chance. One group takes avenciguat tablets and the other group takes placebo tablets. Placebo tablets look like avenciguat tablets but do not contain any medicine. Participants take a tablet twice a day for 8 weeks.

Participants are in the study for 2 to 3 months. During this time, they visit the study site regularly. At 2 of the visits, the doctors check the pressure in the liver vein by inserting a catheter (a long thin tube) that gives information about pressure in the portal vein. The change in blood pressure is then compared between the 2 groups to see whether the treatment works. The doctors also regularly check participants' health and take note of any unwanted effects.

ELIGIBILITY:
Inclusion Criteria:

* Signed and dated written informed consent in accordance with International Council for Harmonisation-Good Clinical Practice (ICH-GCP) and local legislation prior to admission to the trial
* Male or female who is ≥18 (or who is of legal age in countries where that is greater than 18) and ≤75 years old at screening (Visit 1a)
* Diagnosis of cirrhosis due to non-cholestatic liver disease (including Hepatitis C Virus (HCV), Hepatitis B Virus (HBV), Non-Alcoholic Steatohepatitis (NASH), alcohol-related liver disease, autoimmune hepatitis, Wilson's disease, haemachromatosis, alpha-1 antitrypsin (A1At) deficiency)
* One previous clinically significant decompensation event with clinical resolution at least 4 weeks prior start of screening (visit 1a):

  * First variceal haemorrhage
  * First episode of clinically significant ascites (requiring intervention in lifestyle [fluid and salt restriction] or medical treatment)
* Willing and able to undergo Hepatic Venous Pressure Gradient (HVPG) measurements per protocol (based on Investigator judgement)
* If receiving statins must be on a stable dose for at least 3 months prior to screening (Visit 1b), with no planned dose change throughout the trial
* If receiving treatment with Non-Selective Beta-Blocker (NSBBs) or carvedilol must be on a stable dose for at least 1 month prior to screening (Visit 1b), with no planned dose change throughout the trial
* For patient with alcohol-related cirrhosis, abstinence from significant alcohol misuse / abuse for a minimum of 2 months prior to screening (Visit 1a), and the ability to abstain from alcohol throughout the trial (both evaluated based on Investigator judgement)

Further inclusion criteria apply

Exclusion Criteria:

* History of cholestatic chronic liver disease (e.g. primary biliary cholangitis, primary sclerosing cholangitis)
* Trial participants without adequate treatment for HBV, HCV or NASH as per local guidance (e.g. antiviral therapy for chronic HBV or HCV infection or lifestyle modification in NASH)
* If received curative anti-viral therapy for Hepatitis C Virus (HCV), Sustained Virological Response (SVR) sustained for less than 1 years prior to screening
* If receiving anti-viral therapy for HBV, less than 6 months on a stable dose prior to screening, with planned dose change during the trial or HBV DNA detectable
* Weight change ≥5% within 6 months prior screening in patients with NASH
* Must take, or wishes to continue the intake of, restricted concomitant therapy or any concomitant therapy considered likely (based on Investigator judgement) to interfere with the safe conduct of the trial
* Systolic Blood Pressure (SBP) <100 mmHg or Diastolic Blood Pressure (DBP) <70 mmHg at screening (Visit 1a)
* Hepatic impairment defined as a Child-Turcotte-Pugh score ≥8 at screening

Further exclusion criteria apply

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2024-01-03 (Actual); Primary Completion 2024-05-30 (Actual); Study Completion 2024-05-30 (Actual)

CONTACTS AND LOCATIONS:
Locations (15):
- United States (2):
  - California Liver Research Institute, Pasadena, California
  - Inland Empire Clinical Trials, LLC, Rialto, California
- AKH - Medical University of Vienna, Vienna, Austria
- Centre Hospitalier de l'Universite de Montreal (CHUM), Montreal, Quebec, Canada
- China (2):
  - Beijing Friendship Hospital, Beijing
  - NanFang Hosptial, Guangzhou
- France (2):
  - HOP Beaujon, Clichy
  - HOP Rangueil, Toulouse
- Germany (2):
  - Universitätsmedizin der Johannes Gutenberg-Universität Mainz, Mainz
  - Universitätsklinikum Münster, Münster
- Shin-yurigaoka General Hospital, Kanagawa, Kawasaki, Japan
- Regional Institute of Gastroenterology Hepatology "Prof. Dr. O. Fodor", Cluj-Napoca, Romania
- Soon Chun Hyang University Hospital Bucheon, Bucheon-si, Gyeonggi-do, South Korea
- Spain (2):
  - Hospital Vall d'Hebron, Barcelona
  - Hospital Ramón y Cajal, Madrid

IPD SHARING:
Plan to Share IPD: Yes
Once the criteria in section 'time frame frame' are fulfilled , researchers can use the following link https:// www.mystudywindow.com/msw/datasharing to request access to the clinical study documents regarding this study, and upon a signed "Document Sharing Agreement". Furthermore, researchers can request access to the clinical study data, for this and other listed studies, after the submission of a research proposal and according to the terms outlined in the website.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: After structured results have been posted, all regulatory activities are completed in the US and EU for the product and indication, and after the primary manuscript has been accepted for publication.
Access Criteria: For study documents upon signing of a 'Document Sharing Agreement'.For study data 1. after the submission and approval of the research proposal (checks will be performed by the sponsor and/or the independent review panel, including checking that the planned analysis does not compete with sponsor's publication plan); 2. and upon signing of a legal agreement.
URL: https://www.mystudywindow.com/msw/datasharing

REFERENCES:
- See also: Related Info — http://www.mystudywindow.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Multi-national, randomised, double-blind, parallel group, placebo-controlled trial to investigate the safety and tolerability of avenciguat on top of standard of care on portal hypertension. The trial was prematurely discontinued due to the sponsor's decision.
Pre-assignment Details: All participants were screened for eligibility prior to participation in the trial. Participants attended a specialist site which ensured that they (the participants) strictly met all inclusion and none of the exclusion criteria. Participants were not to be allocated to a treatment group if any of the entry criteria were violated.
Period: Overall Study
Arm/Group | Placebo | Avenciguat
Started | 12 | 10
Completed | 0 | 0
Not Completed | 12 | 10
Not completed — Withdrawal by Subject | 0 | 2
Not completed — Study terminated by sponsor | 12 | 8

BASELINE CHARACTERISTICS:
Population: Randomized set (RS): all enrolled trial participants that were entered or randomized to the trial medication.
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Avenciguat | Total
Number analyzed (Participants) | 12 | 10 | 22
Age, Continuous [Mean (Standard Deviation); unit: Years] | 60.3 (10.6) | 59.2 (10.1) | 59.8 (10.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 2 | 7
  Male | 7 | 8 | 15
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 2 | 3
  Not Hispanic or Latino | 11 | 8 | 19
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 3 | 1 | 4
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 9 | 9 | 18
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Hepatic Venous Pressure Gradient (HVPG) [Mean (Standard Deviation); unit: mmHg] | 14.19 (4.49) | 11.55 (3.94) | 12.99 (4.36)

OUTCOME MEASURES:

1. Primary Outcome: Percentage Change in Hepatic Venous Pressure Gradient (HVPG) From Baseline (Measured in mmHg) After 8 Weeks of Treatment
Description: Percentage change in hepatic venous pressure gradient (HVPG) from baseline to Week 8.
Time Frame: At baseline and at Week 8.
Population: As the trial was discontinued prematurely and no patient completed the 8-week treatment period, no data were available to assess the endpoint.
Arm/Group | Placebo | Avenciguat
Number analyzed (Participants) | 0 | 0

2. Secondary Outcome: Occurrence of a Response, Defined as >10% Reduction From Baseline Hepatic Venous Pressure Gradient (HVPG) (Measured in mmHg) After 8 Weeks of Treatment
Description: Occurrence of a response, defined as at least a 10% reduction in the hepatic venous pressure gradient (HVPG) (measured in mmHg) after 8 weeks of treatment.
Time Frame: At baseline and at Week 8.
Population: as for outcome 1
Arm/Group | Placebo | Avenciguat
Number analyzed (Participants) | 0 | 0

3. Secondary Outcome: Occurrence of Further Decompensation Events (Ascites, Variceal Hemorrhage (VH), and / or Overt Hepatic Encephalopathy (HE)) During the 8-week Treatment Period
Description: Number of participants with at least one decompensation events. Ascites, variceal hemorrhage (VH), and hepatic encephalopathy were defined as further decompensations events. As the trial was discontinued prematurely and no patient completed the 8-week treatment period, the data presented reflects the actual on-treatment period.
Time Frame: Up to 46 days.
Population: Treated set (TS): all trial participants who were randomized to the trial medication and were treated with at least one dose.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Avenciguat
Number analyzed (Participants) | 12 | 10
Participants
  Ascites | 0 | 0
  Variceal Hemorrhage | 0 | 0
  Hepatic encephalopathy | 0 | 0

4. Secondary Outcome: Occurrence of CTCAE Grade 3 (or Higher) Hypotension or Syncope Based on Investigator Judgement During the 8-week Treatment Period
Description: Number of participants with grade 3 or higher common terminology criteria for adverse events (CTCAE) hypotension or syncope base on the investigator judgment. As the trial was discontinued prematurely and no patient completed the 8-week treatment period, the data presented reflects the actual on-treatment period.
Time Frame: Up to 46 days.
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Avenciguat
Number analyzed (Participants) | 12 | 10
Participants | 0 | 0

5. Secondary Outcome: Occurrence of Discontinuation Due to Hypotension or Syncope During the 8-week Treatment Period
Description: Number of participants that discontinued avenciguat due to hypotension or syncope. As the trial was discontinued prematurely and no patient completed the 8-week treatment period, the data presented reflects the actual on-treatment period.
Time Frame: Up to 46 days.
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Avenciguat
Number analyzed (Participants) | 12 | 10
Participants | 0 | 0

ADVERSE EVENTS:
Time Frame: All-cause mortality: From first drug administration until individual end of study. Up to 60 days. Adverse event reporting: From first administration until last drug administration plus 7-day residual effect period. Up to 53 days.
Description: Treated set (TS): all trial participants who were randomized to the trial medication and were treated with at least one dose.
Arm/Group | Placebo | Avenciguat
All-Cause Mortality (participants affected / at risk) | 0/12 | 0/10
Serious Adverse Events (participants affected / at risk) | 0/12 | 2/10
Other Adverse Events (participants affected / at risk) | 1/12 | 3/10
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=12) | Avenciguat (N=10)
Sinus arrest (Cardiac disorders) | 0 | 1
Vulval abscess (Infections and infestations) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=12) | Avenciguat (N=10)
Abdominal distension (Gastrointestinal disorders) | 0 | 1
Hyperuricaemia (Metabolism and nutrition disorders) | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Insomnia (Psychiatric disorders) | 1 | 0
Polyuria (Renal and urinary disorders) | 0 | 1
Hypotension (Vascular disorders) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Boehringer Ingelheim (BI) acknowledges that investigators have the right to publish the study results. Investigators shall provide BI with a copy of any publication or presentation for review prior to any submission. Such review will be done with regard to proprietary information, information related to patentable inventions, medical, scientific, and statistical accuracy within 60 days. BI may request a delay of the publication in order to protect BI's intellectual property rights.

DOCUMENTS (2):
  • Study Protocol (2023-11-29): https://cdn.clinicaltrials.gov/large-docs/43/NCT06082843/Prot_000.pdf
  • Statistical Analysis Plan (2024-07-01): https://cdn.clinicaltrials.gov/large-docs/43/NCT06082843/SAP_001.pdf